CLINICAL TRIAL: NCT05979246
Title: A Comparative Prospective Study to Evaluate the Effect of the Superhydrophilic Surface of Lance CLEAR Implants on the Marginal Bone Loss and Survival in Diabetic and Non Diabetic Patients
Brief Title: Effect of the Superhydrophilic Surface of Lance CLEAR Implants on the Marginal Bone Loss and Survival in Diabetic and Non Diabetic Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: MIS Implant Technologies, Ltd (Industry)
Collaborators: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MIS Implants Technologies
Record Dates: First submitted 2023-07-30; First posted 2023-08-07 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-07

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: 40 patients who are planned to undergo implant installation will be enrolled in the study, at the department of Periodontology at the School of postgraduate dentistry in the Rambam Health Care Center.
  The patients will be divided into 2 groups:
  * Test group - 20 patients diagnosed with type 2 diabetes with 10>HbA1C>7.5% values
  * Control group - 20 non-diabetic patients.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Diabetic patients (Experimental): undergo implant installation
  Interventions: Device: Lance CLEAR dental implant

INTERVENTIONS:
Device: Lance CLEAR dental implant — The surgical procedure will be performed by experienced periodontists, all implants will be at least Ø 3.75 mm and 8-11.5 mm long. After reflecting the flaps, a bone biopsy will be harvested as part of the drilling procedure using a Ø 2.4 mm trephine drill and the implants will be seated into a crestal position

SUMMARY:
The aim of this clinical, prospective study involving implants with a superhydrophilic surface is to compare the changes of the peri-implant tissues and the survival rate between diabetics and non-diabetics patients, after 12 months of loading.

hypothesis: It is not expected to find any short-term differences in failures and marginal bone loss between the diabetic and non-diabetic patients. On the longer term higher marginal bone loss may affect the diabetic group 40 patients who are planned to undergo implant installation will be enrolled in the study.

The patients will be divided into 2 groups:

* Test group - 20 patients diagnosed with type 2 diabetes with 10>HbA1C>7.5% values
* Control group - 20 non-diabetic patients.

DETAILED DESCRIPTION:
In recent years, our understanding of the primary processes that affect bone growth around implants has progressed. It was found that the standard surface of most implants is not hydrophilic enough; therefore, it is necessary to increase the healing time to allow sufficient bony apposition at the implant interface, until reaching a satisfactory load-bearing capacity. Studies have demonstrated that surface superhydrophilicity can be gained following storage in an isotonic solution (NaCl); this feature leads to an earlier bone apposition and higher anchorage, already after the very first weeks of implantation.

Hypothesis: It is not expected to find any short-term differences in failures and marginal bone loss between the diabetic and non-diabetic patients. On the longer term higher marginal bone loss may affect the diabetic group.

Aim:to compare the changes of the peri-implant tissues and the survival rate between diabetics and non-diabetics patients, after 12 months of loading.

Methods and Materials: 40 patients who are planned to undergo implant installation will be enrolled in the study, at the department of Periodontology at the School of postgraduate dentistry in the Rambam Health Care Center. .

The patients will be divided into 2 groups:

* Test group - 20 patients diagnosed with type 2 diabetes with 10>HbA1C>7.5% values
* Control group - 20 non-diabetic patients. Visit 0 - Screening Visit 1 - Surgical procedure (± 8 weeks)

After insertion of the implants, the following surgical indicators will be taken:

1. Stability of the implants will be measured using an Osstell device with a fitted peg screwed into the implant neck; unit is given as an arbitrary implant stability quotient (ISQ).
2. Register bone quality type 1-4 according to the doctor report using Bone classification of Lekholm & Zarb ,1985.

Visit 2 - suture removal (10 ±3days) Visit 3 (surgical uncovering) 12 weeks after implantation (±8 weeks) Visit 4 (follow-up) 16 weeks after implantation (± 8 weeks) :this visit includes periodontal examination (PD, BOP, PI, GI) and GCF sampling.

Visit 5 ( Follow up ) 12 months after rehabilitation (± 4 weeks) :Clinical and radiographic assessment of the periimplant mucosa

ELIGIBILITY:
Inclusion Criteria:

1. Ages ≥18.
2. A properly signed and dated consent form.
3. The need to perform a dental implant (up to two dental implants will be selected for the patient).
4. The existence of sufficient alveolar bone that allows the installation of implants of standard size (diameter 3.75 or above and height of at least 8 mm).
5. Patients who will receive a fixed restoration (a crown or three units bridge)
6. A type 2 diabetes with 10 > A1C>7.5 % values but not above 10, or non-diabetic patient (control).
7. Meeting the study schedules and attending the study visits.

Exclusion Criteria:

1. The presence of an active periodontal disease (PD≥6 mm with bleeding on probing).
2. Smoking more than 10 cigarettes a day.
3. Pharmacological condition which can affect the healing of soft or hard tissue.
4. Past radiation therapy to the head and neck.
5. Patients under medications with known effects on bone metabolism (e.g. steroids, anti-TNF-α), antibiotics therapy in the previous months.
6. Impaired occlusion that can lead to pathologies.
7. Pregnancy and lactating.
8. A patient who needs local bone augmentation.
9. Using removable prosthesis in the implantation area.
10. Subjects who are currently enrolled, recently participated (within 30 days prior to screening), or planning to enroll in another study that may conflict with protocol requirements or may confound the subject results in this trial.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
marginal bone loss | one year after loading
  radiographic bone resorption around the implant

SECONDARY OUTCOMES:
Survival rate | 12 weeks after implantation
  Implant stability measurements by Osstell.